CLINICAL TRIAL: NCT02717494
Title: Safety and Immunogenicity of Anti-Pneumococcal Vaccines in HIV-Infected Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD P1091
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: PNC Vaccine; HIV-infected Pregnant Women
Keywords: PPV-23; PCV-10; HIV; Immunization; Pregnancy
MeSH Terms: interventions — 10-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1A (PPV-23) (Experimental): In Step 1, women in Arm 1A were administered a 0.5 milliliter (mL) dose of PPV-23 intramuscularly once.
  Interventions: Biological: PPV-23
- Arm 1B (PCV-10) (Experimental): In Step 1, women in Arm 1B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  Interventions: Biological: PCV-10
- Arm 1C (placebo) (Placebo Comparator): In Step 1, women in Arm 1C were administered a 0.5 mL dose of 0.9 percent Sodium Chloride (NaCl) intramuscularly once.
  Interventions: Other: NaCl
- Arm 2A (PPV-23) (Experimental): In Step 2, women who received placebo in step 1 that were randomized to Arm 2A were administered a 0.5 mL dose of PPV-23 intramuscularly once.
  Interventions: Biological: PPV-23
- Arm 2B (PCV-10) (Experimental): In Step 2, women who received placebo in step 1 that were randomized to Arm 2B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  Interventions: Biological: PCV-10
- Step 3 (PCV-10) (Experimental): In Step 3, women who received placebo in step 1 and failed entry into step 2 due to ongoing new pregnancy were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  Interventions: Biological: PCV-10

INTERVENTIONS:
Biological: PPV-23 — PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
  Arms: Arm 1A (PPV-23); Arm 2A (PPV-23)
Biological: PCV-10 — PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
  Arms: Arm 1B (PCV-10); Arm 2B (PCV-10); Step 3 (PCV-10)
Other: NaCl — NaCl was the placebo for the study against which the two vaccines were compared during pregnancy.
  Arms: Arm 1C (placebo)

SUMMARY:
The purpose of this study was to determine the safety, reactogenicity, immunogenicity, transplacental antibody transfer and interference with infant responses to childhood vaccination of maternal vaccination with pneumococcal conjugate 10-valent vaccine (PCV-10) or pneumococcal polysaccharide 23-valent vaccine (PPV-23) by comparison with placebo.

DETAILED DESCRIPTION:
This was a multi-center, Phase II, randomized, double-blinded, placebo-controlled study of Human Immunodeficiency Virus (HIV)-infected pregnant women on Highly Active Antiretroviral Therapy (HAART) who were in the second or third trimester of pregnancy and of their infants. The study was designed to investigate the safety, reactogenicity, immunogenicity, transplacental antibody transfer and interference with infant responses to childhood vaccination of maternal vaccination with PCV-10 or PPV-23 by comparison with placebo.

Mothers were randomized to one of three arms and received PCV-10, PPV-23, or placebo in a blinded fashion. They were followed for safety, immunogenicity and vaccine-specific anti-capsular pneumococcus (PNC) antibody persistence until 24 weeks post-delivery. Women who received placebo were randomized to a second study step and received PCV-10 or PPV-23 at 24 weeks post-delivery. Antibody responses to the vaccine administered 6 months postpartum were measured. Women who received placebo but cannot be randomized to a second study step due to ongoing new pregnancy were enrolled in a third study step and receive open label PCV-10 at the last study visit; no data were collected on these women and they were not followed after vaccine administration. All infants received PCV-10 vaccinations per local standard of care.

ELIGIBILITY:
Step 1 Inclusion Criteria for Pregnant Women:

1. Pregnant women ≥ 18 years old who provided written informed consent prior to study initiation.
2. Pregnant women < 18 years old with parent or legal guardian able and willing to provide signed informed consent, or who had the capacity to consent for themselves, as defined by the local Institutional Review Board (IRB), and who provided written informed consent prior to study initiation.
3. Gestational age [≥ 14 weeks (14 weeks 0 days) to < 33 weeks (32 weeks 6 days)] documented by the approximate date of the last menstrual period and corroborated by ultrasound if obtained as per local standard of care. Results of the ultrasound were recorded on the Abdominal Ultrasound Form.
4. Documentation of HIV-1 infection defined as positive results from two samples collected at different time points as per standard of care. Results and source documentation may have been obtained from the medical records.
5. Receipt of HAART (a regimen of at least three ARV drugs) for ≥ 4 weeks prior to enrollment.
6. Documented platelet count of > 50,000/mm3 and an absolute neutrophil count (ANC) of > 500/ mm3 ≤ 28 days prior to study entry.
7. Women who were willing and able to comply with the study visits.

Step 1 Exclusion Criteria for Pregnant Women:

1. Receipt of any PCV or PPV-23 at any time prior to enrollment, documented by medical history or record.
2. Receipt of any live licensed vaccine ≤ 4 weeks or inactivated licensed vaccine ≤ 2 weeks prior to study entry.
3. Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) ≤ 4 weeks prior to enrollment in this study, or expectations to receive another non-licensed agent before delivery unless approval from the protocol team is obtained.
4. Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 100.4 degrees F ≤ 24 hours prior to study entry.
5. Women who planed to terminate their pregnancy.
6. Women who had a prior history of lupus or other autoimmune disorders.
7. Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or evidence of immunosuppression as a result of an underlying illness (other than HIV-1 infection) or treatment.
8. Ongoing neoplastic disease (excluding non-melanoma skin cancer, and human papilloma virus-related cervical dysplasia, cervical intraepithelial neoplasia (CIN) grades 1, 2 or 3).
9. Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 12 weeks of study entry.
10. Women who received last dose of corticosteroids for preterm labor ≤ 1 week prior to study entry. Note: A woman can be enrolled if more than 1 week has elapsed from the last dose of corticosteroids, i.e., enrollment may be delayed to satisfy this criterion.
11. Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.
12. Receipt of Interleukin-2 (IL2), interferon (IFN), granulocyte-macrophage colony-stimulating factor (GMCSF) or other immune mediators ≤ 12 weeks before enrollment.
13. History of a severe adverse reaction to inactivated polysaccharide or conjugated vaccines.
14. Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
15. Pregnancy complications (in the current pregnancy) such as pre-term labor, and pre-eclampsia or any other pregnancy related complication, which in the opinion of the investigator might jeopardize the results of the study.
16. Chronic hepatitis B infection that may require administration of Hepatitis B Hyperimmune Globulin to neonates.

Step 2 Inclusion Criteria for Women:

1. 24 weeks ± 4 weeks postpartum.
2. Completion of Step 1.
3. Receipt of placebo on Step 1.

Step 2 Exclusion Criteria for Women:

1. Pregnancy.
2. Receipt of any live licensed vaccine ≤ 4 weeks or inactivated licensed vaccine ≤ 2 weeks prior to Step 2 entry.
3. Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) ≤ 4 weeks prior to vaccination, or expects to receive another non-licensed agent within 28 days after vaccination.
4. Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 100.4 degrees F within 24 hours of entry except when, in the opinion of the physician, withholding the agent entails even greater risk.
5. Use of anti-cancer systemic chemotherapy or radiation therapy or has developed immunosuppression as a result of an underlying illness (other than HIV-1 infection) or treatment.
6. Use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 2 weeks of entry in Step 2.
7. Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) within 12 weeks prior to entry in Step 2 or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during the 28 days following vaccination.
8. Receipt of IL2, IFN, GMCSF or other immune mediators ≤ 12 weeks before entry in Step 2.

Step 3 Inclusion Criteria for Women

1. 24 weeks ± 4 weeks postpartum.
2. Completion of Step 1.
3. Receipt of placebo on Step 1.
4. Met Step 2 exclusion criterion of pregnancy.

Step 3 Exclusion Criteria for Women

None.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Study Chair — University of Colorado, Denver; Marisa Mussi, MD, Study Chair — University of Sao Paulo Ribeirão Preto School of Medicine; Geraldo Duarte, MD, Study Chair — University of Sao Paulo Ribeirão Preto School of Medicine
Locations (8):
- Brazil (8):
  - FUNDEP (Belo Horizonte), Belo Horizonte, Minas Gerais
  - Hospital Geral de Nova Iguaçu Avenida Henrique Duque Estrada Mayer, Nova Iguaçu, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteria, Rio de Janeiro, Rio de Janeiro
  - Hospital dos Servidores (Rio de Janeiro), Saúde, Rio de Janeiro
  - Universidade de Caxias do Sul. Brasil, Caxias do Sul, Rio Grande do Sul
  - Hospital Santa Casa Porto Alegre Brazil, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Ribeirão Preto Medical School, University of São Paulo, Brazil, Ribeirão Preto, São Paulo

REFERENCES:
- [Derived] Duarte G, Muresan P, Ward S, Laimon L, Pelton SI, Canniff J, Golner A, Bone F, Newton L, Fenton T, Coutinho CM, Joao EC, Santos BR, Pilotto JH, Oliveira RH, Pinto JA, Machado ES, Kreitchman R, Chakhtoura N, Mussi-Pinhata MM, Weinberg A. Immunogenicity of Conjugated and Polysaccharide Pneumococcal Vaccines Administered During Pregnancy or Postpartum to Women With HIV. J Infect Dis. 2022 Mar 15;225(6):1021-1031. doi: 10.1093/infdis/jiab567. PMID 34791324
- [Derived] Weinberg A, Muresan P, Laimon L, Pelton SI, Goldblatt D, Canniff J, Zimmer B, Bone F, Newton L, Fenton T, Kiely J, Johnson MJ, Joao EC, Santos BR, Machado ES, Pinto JA, Chakhtoura N, Duarte G, Mussi-Pinhata MM; NICHD P1091 study team. Safety, immunogenicity, and transplacental antibody transport of conjugated and polysaccharide pneumococcal vaccines administered to pregnant women with HIV: a multicentre randomised controlled trial. Lancet HIV. 2021 Jul;8(7):e408-e419. doi: 10.1016/S2352-3018(20)30339-8. Epub 2021 Apr 27. PMID 33915104
- See also: NICHD website — https://www.nichdclinicalstudies.org/
- See also: The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from April 2016 to November 2017. Participants were recruited from medical clinics.
Pre-assignment Details: Of the 347 pregnant women enrolled in the study, 346 were randomized and received study vaccination. One discontinued study prior to receiving study vaccination.
  There were 349 infants born on the study, including 4 sets of twins. Two women discontinued study prior to delivering their child. Those children are not included in the outcome results.
Period: First Intervention (Step 1)
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Started | 115 | 115 | 116
Were Randomized to Step 2A (PPV-23) (Women who received Placebo in Step 1, and were randomized to Step 2A to receive PPV-23.) | 0 | 0 | 53
Were Randomized to Step 2B (PCV-10) (Women who received Placebo in Step 1, and were randomized to Step 2B to receive PCV-10.) | 0 | 0 | 53
Were Enrolled in Step 3 (PCV-10) (Women who received Placebo in Step 1 but were pregnant again, enrolled in Step 3.) | 0 | 0 | 4
Completed | 109 | 108 | 111
Not Completed | 6 | 7 | 5
Not completed — Lost to Follow-up | 4 | 7 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Death | 0 | 0 | 1
Period: Second Intervention (Step 2 or Step 3)
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Started | 0 (Only Step 1 placebo recipients were enrolled in Step 2.) | 0 (Only Step 1 placebo recipients were enrolled in Step 2.) | 110 (One participant who completed Step 1 did not enroll in Step 2.)
Completed Step 2A | 0 | 0 | 52
Completed Step 2B | 0 | 0 | 50
Completed Step 3 | 0 | 0 | 4
Completed | 0 | 0 | 106
Not Completed | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Mother participants who received study treatment in Step 1 were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo) | Total
Number analyzed (Participants) | 115 | 115 | 116 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] — This is age at randomization, in years.
  years | 28 (6) | 27 (6) | 28 (6) | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 115 | 116 | 346
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110 | 112 | 113 | 335
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 4 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 57 | 51 | 61 | 169
  White | 19 | 24 | 25 | 68
  More than one race | 36 | 40 | 28 | 104
  Unknown or Not Reported | 3 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Brazil | 115 | 115 | 116 | 346
Gestational Age at Randomization [Mean (Standard Deviation); unit: weeks] — This is the estimated gestational age at study randomization, in weeks.
  weeks | 25 (5) | 25 (5) | 26 (5) | 26 (5)
CD4% at Randomization [Mean (Standard Deviation); unit: percent] | 32 (9) | 32 (9) | 31 (9) | 32 (9)
CD4 Count at Randomization [Mean (Standard Deviation); unit: cells/microliter] | 585 (257) | 596 (243) | 564 (297) | 582 (266)
RNA Copies at Randomization [Mean (Standard Deviation); unit: copies/mL] | 569 (1825) | 307 (1278) | 1144 (7864) | 674 (4730)
Log10 RNA Copies at Randomization [Mean (Standard Deviation); unit: log10(copies)/mL] | 1.9 (0.6) | 1.9 (0.5) | 1.8 (0.6) | 1.9 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Experienced Various Adverse Events (AEs)
Description: The number of women who experienced grade ≥ 3 adverse events (AEs) in the 4 weeks after vaccination in Step 1 and grade 4 AEs or death up to 24 weeks post-partum. AE grading (Grade 1- mild to Grade 4-life-threatening) was done by DAIDS AE Grading table v2.0 (see References).
Time Frame: up to 24 Weeks Post-Delivery for mother participants.
Population: All women randomized to vaccine or placebo, and who received the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Number analyzed (Participants) | 115 | 115 | 116
Participants
  Grade 3+ AEs, up to week 4, Step 1 | 2 | 3 | 4
  Grade 4+ AEs, after week 4, Step 1 | 1 | 2 | 4
  Grade 3+ AEs related to treatment, Step 1 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Arm 1A (PPV-23); Test type: Other; % with grade 3+ AEs, up to week 4 Step 1 = 2, 90% CI 2-sided [0 to 5] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Arm 1B (PCV-10); Test type: Other; % with grade 3+ AEs, up to week 4 Step 1 = 3, 90% CI 2-sided [1 to 7] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 3: Comparison: Arm 1C (Placebo); Test type: Other; % with grade 3+ AEs up to week 4, Step 1 = 3, 90% CI 2-sided [1 to 8] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 4: Comparison: Arm 1A (PPV-23); Test type: Other; % with grade 4+ AEs after week 4, Step 1 = 1, 90% CI 2-sided [0 to 4] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 5: Comparison: Arm 1B (PCV-10); Test type: Other; % with grade 4+ AEs after week 4, Step 1 = 2, 90% CI 2-sided [0 to 5]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 6: Comparison: Arm 1C (Placebo); Test type: Other; % with grade 4+ AEs, after week 4 Step 1 = 3, 90% CI 2-sided [1 to 8] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 7: Comparison: Arm 1A (PPV-23); Test type: Other; % with Grade 3+ related to treatment = 1, 90% CI 2-sided [0 to 4] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 8: Comparison: Arm 1B (PCV-10); Test type: Other; % with Grade 3+ related to treatment = 1, 90% CI 2-sided [0 to 4] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 9: Comparison: Arm 1C (Placebo); Test type: Other; % with Grade 3+ related to treatment = 1, 90% CI 2-sided [0 to 4] — Confidence intervals were Exact Clopper-Pearson

2. Primary Outcome: Number of Women Who Experienced Grade ≥ 3 Adverse Events (AEs) in Step 2
Description: The number of women who enrolled in Step 2, received vaccine and who experience grade ≥ 3 adverse events (AEs) in the 4 weeks after vaccination in Step 2 is presented.
Time Frame: up to 4 Weeks after Step 2 vaccination for Mother Participants
Population: Women who received Placebo in Step 1 and who were eligible and were randomized to Step 2.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2A (PPV-23): In Step 2, women who received Placebo in Step 1 and who were randomized to Arm 2A were administered a 0.5 mL dose of PPV-23 intramuscularly once.
  PPV-23: PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
- Arm 2B (PCV-10): In Step 2, women who received Placebo in Step 1 and who were randomized to Arm 2B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  PCV-10: PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
Arm/Group | Arm 2A (PPV-23) | Arm 2B (PCV-10)
Number analyzed (Participants) | 53 | 53
Participants
  Grade 3+ AEs, up to week 4, Step 2 | 0 | 0
  Grade 3+ AEs related to treatment, Step 2 | 0 | 0
Statistical Analysis 1: Comparison: Arm 2A (PPV-23); Test type: Other; % with grade 3+ AEs, up to week 4 Step 2 = 0, 90% CI 2-sided [0 to 5] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Arm 2B (PCV-10); Test type: Other; % with grade 3+ AEs, up to week 4 Step 2 = 0, 90% CI 2-sided [0 to 5] — Confidence intervals were Exact Clopper-Pearson

3. Primary Outcome: Number of Infants With Various Adverse Events Following Maternal Vaccination With PCV10 and PPV23 Administered in Pregnancy
Description: The number of infants who experience grade ≥ 3 adverse events (AEs), congenital defects, HIV infections or pneumonia, meningitis or IPD after maternal vaccination in Step 1, assessed from birth through 24 weeks of life for infant participants.
Time Frame: through 24 weeks of life for infant participants
Population: Infants who were born on the study.
Measure: Count of Participants; unit: Participants
Groups:
- Infants Born to Women in Arm 1A (PPV-23): In Step 1, women in Arm 1A were administered a 0.5 milliliter (mL) dose of PPV-23 intramuscularly once.
  PPV-23: PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
- Infants Born to Women in Arm 1B (PCV-10): In Step 1, women in Arm 1B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  PCV-10: PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
- Infants Born to Women in Arm 1C (Placebo): In Step 1, women in Arm 1C were administered a 0.5 mL dose of 0.9 percent Sodium Chloride (NaCl) intramuscularly once.
  NaCl: NaCl was the placebo for the study against which the two vaccines were compared during pregnancy.
Arm/Group | Infants Born to Women in Arm 1A (PPV-23) | Infants Born to Women in Arm 1B (PCV-10) | Infants Born to Women in Arm 1C (Placebo)
Number analyzed (Participants) | 112 | 116 | 119
Participants
  Grade 3+ AEs, | 23 | 23 | 24
  Congenital Anomalies | 19 | 25 | 15
  HIV Infected | 0 | 0 | 0
  Pneumonia, meningitis or IPD | 5 | 8 | 8
Statistical Analysis 1: Comparison: Infants Born to Women in Arm 1A (PPV-23); Test type: Other; % infants with grade 3+ AEs = 21, 90% CI 2-sided [14 to 28] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Infants Born to Women in Arm 1B (PCV-10); Test type: Other; % infants with grade 3+ AEs = 20, 90% CI 2-sided [14 to 27]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 3: Comparison: Infants Born to Women in Arm 1C (Placebo); Test type: Other; % infants with grade 3+ AEs = 20, 90% CI 2-sided [14 to 27] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 4: Comparison: Infants Born to Women in Arm 1A (PPV-23); Test type: Other; % infants with congenital anomalies = 17, 90% CI 2-sided [11 to 24]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 5: Comparison: Infants Born to Women in Arm 1B (PCV-10); Test type: Other; % infants with congenital anomalies = 22, 90% CI 2-sided [15 to 29]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 6: Comparison: Infants Born to Women in Arm 1C (Placebo); Test type: Other; % infants with congenital anomalies = 13, 90% CI 2-sided [8 to 19] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 7: Comparison: Infants Born to Women in Arm 1A (PPV-23); Test type: Other; % infants with HIV infection = 0, 90% CI 2-sided [0 to 3]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 8: Comparison: Infants Born to Women in Arm 1B (PCV-10); Test type: Other; % infants with HIV infection = 0, 90% CI 2-sided [0 to 3] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 9: Comparison: Infants Born to Women in Arm 1C (Placebo); Test type: Other; % infants with HIV infection = 0, 90% CI 2-sided [0 to 2] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 10: Comparison: Infants Born to Women in Arm 1A (PPV-23); Test type: Other; % with pneumonia, meningitis or IPD = 4, 90% CI 2-sided [2 to 9] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 11: Comparison: Infants Born to Women in Arm 1B (PCV-10); Test type: Other; % with pneumonia, meningitis or IPD = 7, 90% CI 2-sided [3 to 12] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 12: Comparison: Infants Born to Women in Arm 1C (Placebo); Test type: Other; % with pneumonia, meningitis or IPD = 7, 90% CI 2-sided [3 to 12] — Confidence intervals were Exact Clopper-Pearson

4. Primary Outcome: Number of Women With a Two-fold or Higher Increase in ELISA-measured IgG PNC Antibody Concentrations
Description: The number of participants with a two-fold or higher increase in ELISA-measured IgG PNC antibody concentrations from baseline to 28 days after immunization in Step 1 to 1 or more serotypes.
  The proportion of participants with >=0.35ug/mL ELISA-measured IgG PNC antibody concentrations at 28 days after immunization in Step 1 to 1 or more serotypes.
Time Frame: 28 days after Immunization in Step 1
Population: Pregnant women who received the vaccination and did not deliver prior to the day 28 study visit and who had ELISA-measured IgG PNC antibody concentrations measured at baseline and at 28 days after immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Number analyzed (Participants) | 110 | 114 | 113
Participants
  >=2 fold change from baseline to day 28 | 106 | 112 | 7
  >=0.35ug.mL at day 28 | 109 | 114 | 106
Statistical Analysis 1: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority — This is the test to compare the two vaccine arms with respect to proportion of participants with >=2 fold increase at day 28; p = 0.44, Fisher Exact — The threshold for statistical significance is 0.05; Fisher's exact test was used because 50% of the cells had expected counts less than 5
Statistical Analysis 2: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority — This is the test to compare the two vaccine arms with respect to proportion of participants with values >=0.35ug/mL at day 28; p = 0.49, Fisher Exact — The threshold for statistical significance is 0.05; Fisher's exact test was used because 50% of the cells had expected counts less than 5
Statistical Analysis 3: Comparison: Arm 1A (PPV-23); Test type: Other; % vaccinees with >=2fold increase = 96, 95% CI 2-sided [91 to 99] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 4: Comparison: Arm 1B (PCV-10); Test type: Other; % vaccinees with >=2fold increase = 98, 95% CI 2-sided [94 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 5: Comparison: Arm 1C (Placebo); Test type: Other; % with >=2 fold increase = 6, 95% CI 2-sided [3 to 12] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 6: Comparison: Arm 1A (PPV-23); Test type: Other; % vaccinees with >=0.35ug/mL at day 28 = 99, 95% CI 2-sided [95 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 7: Comparison: Arm 1B (PCV-10); Test type: Other; % vaccinees with >=0.35ug/mL at day 28 = 100, 95% CI 2-sided [97 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 8: Comparison: Arm 1C (Placebo); Test type: Other; % with >=0.35ug/mL at day 28 = 94, 95% CI 2-sided [88 to 97] — Confidence intervals were Exact Clopper-Pearson

5. Primary Outcome: Number of Infant Participants With ELISA-measured IgG PNC Antibody Levels ≥ 0.35ug/mL at 8 Weeks of Age
Description: The number of infant participants with ELISA-measured IgG PNC antibody levels ≥ 0.35ug/mL at 8 weeks of age to 1 or more serotypes.
Time Frame: 8 Weeks of Life
Population: The are the infants who were born on study and who had blood drawn for the week 8 evaluation prior to receiving their PCV-10 vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1A (PPV-23): These are the infants born to the pregnant women in Arm 1A. In Step 1, women in Arm 1A were administered a 0.5 milliliter (mL) dose of PPV-23 intramuscularly once.
  PPV-23: PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
- Arm 1B (PCV-10): These are the infants born to the pregnant women in Arm 1B. In Step 1, women in Arm 1B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  PCV-10: PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
- Arm 1C (Placebo): These are the infants born to women enrolled in Arm 1C. In Step 1, women in Arm 1C were administered a 0.5 mL dose of 0.9 percent Sodium Chloride (NaCl) intramuscularly once.
  NaCl: NaCl was the placebo for the study against which the two vaccines were compared during pregnancy.
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Number analyzed (Participants) | 105 | 108 | 109
Participants | 87 | 95 | 46
Statistical Analysis 1: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority; p = 0.29, Chi-squared — The threshold for statistical significance is 0.05

6. Secondary Outcome: Ratio of Infant/Mother PNC Antibody Levels
Description: The ratios of infant/mother PNC antibody levels to study used serotypes.
Time Frame: At Delivery for Mother Participants and Birth for Infant Participants
Population: These are the mother-infant pairs who meet the criteria of receipt of study product for the moms and have data for delivery/birth time point.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Number analyzed (Participants) | 109 | 113 | 115
ratio | 0.92 [0.91 to 0.93] | 0.93 [0.92 to 0.94] | 0.90 [0.89 to 0.91]
Statistical Analysis 1: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority; p = 0.08, t-test, 2 sided — The threshold for statistical significance is 0.05

7. Secondary Outcome: Number of Participants With a >=0.35ug/mL ELISA-measured IgG PNC Antibody Concentrations at Labor/Delivery and 24 Weeks Post-partum
Description: The number of participants with a >=0.35ug/mL ELISA-measured IgG PNC antibody concentrations at the time points listed for 1 or more serotypes.
Time Frame: at Labor and Delivery and 24 Weeks Post-Delivery for Mother Participants
Population: Pregnant women who received the vaccination and did not deliver prior to the day 28 study visit and who had ELISA-measured IgG PNC antibody concentrations measured at the timepoints listed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo)
Number analyzed (Participants) | 113 | 115 | 116
Participants
  at labor and delivery | 109 | 115 | 16
  at 24 weeks post partum: number analyzed (Participants) | 107 | 108 | 105
  at 24 weeks post partum | 105 | 107 | 58
Statistical Analysis 1: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority — This is the test to compare the two vaccine arms with respect to proportion of participants with >=2 fold increase at labor and delivery; p = 0.37, Chi-squared — The threshold for statistical significance is 0.05
Statistical Analysis 2: Comparison: Arm 1A (PPV-23) vs Arm 1B (PCV-10); Test type: Superiority — This is the test to compare the two vaccine arms with respect to proportion of participants with >=2 fold increase at 24 weeks post partum; p = 0.21, Fisher Exact; Fisher's exact test was used because 50% of the cells had expected counts less than 5

8. Secondary Outcome: Number of Participants With a Two-fold or Higher Increase in ELISA-measured IgG PNC Antibody Concentrations at 28 Days After PPV-23 Vaccination in Step 1 and Step 2
Description: The number of participants with a two-fold or higher increase in ELISA-measured IgG PNC antibody concentrations from baseline to 28 days after immunization in Step 1 vs from entry to Step 2 to 28 days after immunization in Step 2 to 1 or more serotypes.
Time Frame: 28 days after Immunization in Step 1 and in Step 2
Population: Women who received PPV-23 in Step 1 or in Step 2 and who had ELISA-measured IgG PNC antibody concentrations data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A (PPV-23) | Arm 2A (PPV-23)
Number analyzed (Participants) | 110 | 51
Participants | 106 | 49
Statistical Analysis 1: Comparison: Arm 1A (PPV-23); Test type: Other; The threshold for statistical significance is 0.05; % vaccinees with >=2fold increase = 96, 95% CI 2-sided [91 to 99] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Arm 2A (PPV-23); Test type: Other; % vaccinees with >=2fold increase = 98, 95% CI 2-sided [89 to 100] — Confidence intervals were Exact Clopper-Pearson

9. Secondary Outcome: Number of Participants With a Two-fold or Higher Increase in ELISA-measured IgG PNC Antibody Concentrations at 28 Days After PCV-10 Vaccination in Step 1 and Step 2
Description: The proportion of participants with a two-fold or higher increase in ELISA-measured IgG PNC antibody concentrations from baseline to 28 days after immunization in Step 1 vs from entry to Step 2 to 28 days after immunization in Step 2 to 1 or more serotypes.
Time Frame: 28 days after Immunization in Step 1 and in Step 2
Population: Women who received PCV-10 in Step 1 or in Step 2 and who had ELISA-measured IgG PNC antibody concentrations data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1B (PCV-10) | Arm 2B (PCV-10)
Number analyzed (Participants) | 114 | 48
Participants | 112 | 48
Statistical Analysis 1: Comparison: Arm 1B (PCV-10); Test type: Other; % vaccinees with >=2fold increase = 98, 95% CI 2-sided [94 to 100]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Arm 2B (PCV-10); Test type: Other; % vaccinees with >=2fold increase = 100, 95% CI 2-sided [93 to 100] — Confidence intervals were Exact Clopper-Pearson

10. Secondary Outcome: Number of Infant Participants With ELISA-measured IgG PNC Antibody Levels ≥ 0.35ug/mL at 16 and 24 Weeks of Age
Description: The number of infant participants with ELISA-measured IgG PNC antibody levels ≥ 0.35ug/mL at 16 and 24 weeks of age to 1 or more serotypes.
Time Frame: at weeks 16 and 24 of life
Population: These are the infants who were born on study and received the PCV-10 vaccination in the windows allowed by the protocol (prior to week 8 and prior to week 16). The number of infants with nonmissing data who received the vaccination as required are indicated.
Measure: Count of Participants; unit: Participants
Groups:
- Infants of Mothers in Arm 1A (PPV-23): These are the infants born to women enrolled in Arm 1A. In Step 1, women in Arm 1A were administered a 0.5 milliliter (mL) dose of PPV-23 intramuscularly once.
  PPV-23: PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
- Infants of Mothers in Arm 1B (PCV-10): These are the infants born to women enrolled in Arm 1B. In Step 1, women in Arm 1B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  PCV-10: PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
- Infants of Mothers in Arm 1C (Placebo): These are the infants born to women enrolled in Arm 1C. In Step 1, women in Arm 1C were administered a 0.5 mL dose of 0.9 percent Sodium Chloride (NaCl) intramuscularly once.
  NaCl: NaCl was the placebo for the study against which the two vaccines were compared during pregnancy.
Arm/Group | Infants of Mothers in Arm 1A (PPV-23) | Infants of Mothers in Arm 1B (PCV-10) | Infants of Mothers in Arm 1C (Placebo)
Number analyzed (Participants) | 102 | 99 | 99
Participants
  at week 16: number analyzed (Participants) | 100 | 96 | 98
  at week 16 | 100 | 94 | 95
  at week 24 | 102 | 98 | 97
Statistical Analysis 1: Comparison: Infants of Mothers in Arm 1A (PPV-23); Test type: Other; % infants with >=0.35ug/mL at week 16 = 100, 95% CI 2-sided [96 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 2: Comparison: Infants of Mothers in Arm 1B (PCV-10); Test type: Other; % infants with >=0.35ug/mL at week 16 = 98, 95% CI 2-sided [93 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 3: Comparison: Infants of Mothers in Arm 1C (Placebo); Test type: Other; % infants with >=0.35ug/mL at week 16 = 97, 95% CI 2-sided [91 to 99]; Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 4: Comparison: Infants of Mothers in Arm 1A (PPV-23); Test type: Other; % infants with >=0.35ug/mL at week 24 = 100, 95% CI 2-sided [96 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 5: Comparison: Infants of Mothers in Arm 1B (PCV-10); Test type: Other; % infants with >=0.35ug/mL at week 24 = 99, 95% CI 2-sided [95 to 100] — Confidence intervals were Exact Clopper-Pearson
Statistical Analysis 6: Comparison: Infants of Mothers in Arm 1C (Placebo); Test type: Other; % infants with >=0.35ug/mL at week 24 = 98, 95% CI 2-sided [93 to 100] — Confidence intervals were Exact Clopper-Pearson

ADVERSE EVENTS:
Time Frame: For women: up to 28 weeks post-delivery (24 weeks +4 week window) for Steps 1A, 1B, 1C or those who continued to Step 3 (no additional safety follow-up was performed in Step 3); 4 weeks for Steps 2A and 2B; and up to 28 weeks for infants (24 weeks +4 week window).
Description: For women: all grade >=2 signs/symptoms and diagnoses, and all hematology (CBC with differential and platelet count) adverse events. AEs collected for infants: infant death, congenital anomalies, prematurity, low birth weight, neonatal infections/sepsis, Neonatal Intensive Care Unit (NICU) admission, HIV transmission to infant, functional defects (hearing impairment, growth impairment, developmental delay) and Grade ≥ 3 AEs. SAEs were reported according to DAIDS EAE Manual V2.0 (see References).
Groups:
- Arm 2A (PPV-23): In Step 2, women in Arm 2A were administered a 0.5 milliliter (mL) dose of PPV-23 intramuscularly once.
  PPV-23: PPV-23 was a polysaccharide PNC vaccine, licensed in Brazil, directed against 23 serotypes.
- Arm 2B (PCV-10): In Step 2, women in Arm 2B were administered a 0.5 mL dose of PCV-10 intramuscularly once.
  PCV-10: PCV-10 was a conjugate PNC vaccine, licensed in Brazil, directed against 10 serotypes.
Arm/Group | Arm 1A (PPV-23) | Arm 1B (PCV-10) | Arm 1C (Placebo) | Arm 2A (PPV-23) | Arm 2B (PCV-10) | Infants of Mothers in Arm 1A (PPV-23) | Infants of Mothers in Arm 1B (PCV-10) | Infants of Mothers in Arm 1C (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115 | 1/116 | 0/53 | 0/53 | 1/114 | 1/116 | 0/119
Serious Adverse Events (participants affected / at risk) | 15/115 | 15/115 | 16/116 | 0/53 | 0/53 | 20/114 | 21/116 | 19/119
Other Adverse Events (participants affected / at risk) | 66/115 | 63/115 | 62/116 | 5/53 | 7/53 | 9/115 | 8/117 | 17/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1A (PPV-23) (N=115) | Arm 1B (PCV-10) (N=115) | Arm 1C (Placebo) (N=116) | Arm 2A (PPV-23) (N=53) | Arm 2B (PCV-10) (N=53) | Infants of Mothers in Arm 1A (PPV-23) (N=114) | Infants of Mothers in Arm 1B (PCV-10) (N=116) | Infants of Mothers in Arm 1C (Placebo) (N=119)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Uterine infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foetal distress syndrom (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 6 | 5 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Preterm premature rupture (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congenital hydrocephalus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fever neonatal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 5
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | NA | NA | 2 | 2 | 2
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | NA | NA | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | NA | NA | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | NA | NA | 1 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | NA | NA | 0 | 0 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | NA | NA | 1 | 1 | 1
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | NA | NA | 0 | 0 | 1
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 0 | 1 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 0 | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 1 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 1 | 1 | 0
Transient tachypnoea of newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 1 | 2 | 1
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | NA | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | NA | NA | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1A (PPV-23) (N=115) | Arm 1B (PCV-10) (N=115) | Arm 1C (Placebo) (N=116) | Arm 2A (PPV-23) (N=53) | Arm 2B (PCV-10) (N=53) | Infants of Mothers in Arm 1A (PPV-23) (N=115) | Infants of Mothers in Arm 1B (PCV-10) (N=117) | Infants of Mothers in Arm 1C (Placebo) (N=119)
Abdominal pain (Gastrointestinal disorders) | 14 | 18 | 5 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 10 | 5 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 3 | 13 | 1 | 3 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 8 | 9 | 5 | 1 | 2 | 5 | 5 | 8
Urinary tract infection (Infections and infestations) | 3 | 0 | 8 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 5 | 7 | 12 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 6 | 8 | 7 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 38 | 32 | 29 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 18 | 11 | 18 | 1 | 2 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 8 | 9 | 10 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02717494/SAP_000.pdf
  • Study Protocol (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02717494/Prot_001.pdf